CLINICAL TRIAL: NCT06356220
Title: GF-NOURISH (Gluten Free Nutrition Optimization Through Ultra-processed Food Reduction and Improved Strategies for Health)
Acronym: GF-NOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nan Du, Instructor, Attending, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00046867
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Celiac Disease in Children; Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: 1. Study Design: Prospective randomized controlled trial.
  2. Study population: Children (N=120) with newly diagnosed CeD
  3. Intervention: Gluten-Free Food Guide, a nutritional education program focused on minimizing ultra-processed foods in gluten-free die(GFFG), OR a conventional GFD nutritional education class. The nutrition educational program will be based on validated GFD education program. The investigators will use a randomized control trial to assess improvement of overall diet quality, changes in body composition, and minimize toxic and nutrient metal exposures associated with processed gluten-free foods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GFFG (Experimental): Our Canadian collaborators have created Gluten Free-Food Guide (GFFG), a validated nutritional educational intervention, which targets increasing consumption of natural gluten free foods and limiting UPFs. However, this intervention has not yet been applied to a pediatric cohort in the United States. Preliminary data demonstrate enrollment feasibility and generalizability of the intervention. The GFFG arm will have increased focus on plant proteins, minimally processed food intake and fruit/vegetable intake with emphasis on naturally gluten-free foods. The GFFG class will highlight that not all gluten-free foods have the same nutritional and health benefits.
  Interventions: Other: Gluten-Free Diet Education
- Conventional GFD Nutrition Education (Active Comparator): Diet counselling in both the conventional GFD nutrition education and the GFFG intervention arm will include concepts related to nutrition literacy (food label reading, gluten identification, nutritional adequacy). The control group will be provided with the GFFG at the end of the study.
  Interventions: Other: Gluten-Free Diet Education

INTERVENTIONS:
Other: Gluten-Free Diet Education — The two groups will receive different gluten free diet education interventions. Currently, virtual GFD education classes are the standard of care for educating children with CeD and their families about GFD at Boston Children's Hospital. Thus, all diet education (including GFFG intervention) will be provided virtually by Registered Dietitians with expertise in GFDs. .

SUMMARY:
The investigators propose the Gluten Free Nutrition Optimization through Ultra-processed food Reduction and Improved Strategies for Health (GF-NOURISH) study to demonstrate the feasibility and success of a nutritional education program focused on naturally occurring gluten-free foods and minimizing ultra-processed gluten-free foods. The investigators hypothesize that nutritional educational (GF-NOURISH) intervention will have multiple health benefits

DETAILED DESCRIPTION:
Celiac Disease (CeD) is a gluten driven enteropathy that affects up to 3% of the population and typically develops in childhood. Lifelong adherence to a gluten-free diet (GFD) is the primary treatment. Rice, the most common gluten-free substitute grain, naturally bioaccumulates inorganic arsenic. Chronic arsenic exposure may affect neurodevelopment, increase risk of cardiovascular disease and cause kidney damage. In a prior prospective cohort study, the investigators demonstrated that urine arsenic levels increased 2-3 times in newly diagnosed children 6 months after adoption of a GFD. This likely is a consequence of both impaired absorption of vitamin B12 and folate in the small intestine (both nutrients are part of the pathway to excrete arsenic from the body) and increased ingestion of rice products on a gluten-free diet. In particular, gluten-free ultra-processed free foods tend to be specialty products that are made predominantly from rice products, easy for families to identify as safe when avoiding gluten, and rarely fortified with vitamins. Ultra-processed food(UPF) consumption has also been associated with lower perceived quality of life in patients with CeD.

Given the risks associated with gluten-free ultra-processed food, the investigators propose the Gluten Free Nutrition Optimization through Ultra-processed food Reduction and Improved Strategies for Health (GF-NOURISH) study to demonstrate the feasibility and success of a nutritional education program focused on naturally occurring gluten-free foods and minimizing ultra-processed gluten-free foods. The investigators hypothesize that nutritional educational (GF-NOURISH) intervention will have multiple health benefits

The investigators propose to randomize (1:1) 120 children at celiac disease diagnosis to either a novel nutritional education (GF-NOURISH) focused on minimizing ultra-processed gluten free foods or to a conventional GFD nutritional education. Urine/Hair/Toenail arsenic, changes in percent fat free mass, household budgets, diet quality measurements will be evaluated after 6 months on the GFD.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-18 years of age with recent celiac disease diagnosis

Exclusion Criteria:

* Allergic to <3 of the top 8 food allergens
* Co-morbid conditions treated with dietary modifications or that influence nail arsenic values

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of GFFG versus conventional GFD class on body composition, specifically fat free mass | Over 6 months
  While the gold standard measurement for body composition is dual energy X-ray absorptiometry (DEXA) or underwater weighing and air displacement plethysmography (BodPod), these techniques require special facilities that increase cost, are difficult to perform in outpatient settings. DEXA scans also involve radiation exposure. Therefore, the investigators will use bio-impedance spectroscopy analysis (BSA), which is a simple, noninvasive, reproducible, portable and convenient method to measure body composition.26 BSA utilizes body resistance and reactance to derive phase angle (PhA) and estimate the fat (FM) and non-fat (FFM) components of the body

SECONDARY OUTCOMES:
To compare the effect of GFFG vs conventional GFD class on diet quality | Over 6 months
  Given that one of primary objectives of the GFFG is to decrease ultra-processed gluten-free foods (UPGFF), this aim focuses on assessing the impact of the nutrition education intervention on participant's recorded UPF consumption and diet quality. All participants will fill out a three-day food frequency record at study entry and six months of GFD. Food items will be classified by the NOVA system: the most used identification system for UPFs. Of the four leading food processing-based classification systems (NOVA, IARC(International Agency for Research on Cancer), IFIC(International Food Information Council) and UNC(University of North Carolina)), NOVA has been used in 95% of studies on consumption of highly processed foods and chronic health outcome published between 2015 and 2019 in children and adults. NOVA categorizes all the foods by level of food processing: i) unprocessed or minimally processed, (ii) processed culinary ingredients, (iii) processed foods and (iv) UPFs.
To compare the effect of GFFG versus conventional GFD on arsenic exposure | Over 6 months
  The outcome is nail arsenic level after six months on GFD. Toenails will be stored at room temperature and are stable as heavy metals naturally bind to keratin. Toenails will be cleaned to remove exogenous contamination, and then, acid digested.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No